CLINICAL TRIAL: NCT06965582
Title: A Pilot Study Of The ALPFA Benign Prostatic Hyperplasia (BPH) Pulsed Field Ablation (PFA) System In Men With Symptomatic Benign Prostatic Hyperplasia
Brief Title: A Pilot Study Of The ALPFA Benign Prostatic Hyperplasia (BPH) Pulsed Field Ablation (PFA) System
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: ALPFA Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-00001
Record Dates: First submitted 2025-04-27; First posted 2025-05-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: ALPFA BPH PFA System

INTERVENTIONS:
Device: ALPFA BPH PFA System — PFA system for treatment of Benign Prostatic Hyperplasia

SUMMARY:
The ALPFA Medical BPH Pilot Study is a prospective, open label, single arm pilot study to assess the use of the ALPFA BPH PFA System in the treatment of men over the age of 45 with obstructive urinary symptoms associated with BPH.

Male subjects will be consented and undergo protocol-defined baseline assessments. Those who meet study entry criteria will be enrolled and treated with the ALPFA BPH PFA System and then undergo follow-up with protocol-defined assessment.

ELIGIBILITY:
Inclusion:

1. Patients who are ≥ 45 years of age on the day of enrollment.
2. Patients who have failed to achieve satisfactory resolution of BPH symptoms using an approved medication.
3. Life expectancy: the patient has a life expectancy of ≥ 1 year
4. Patient participation: The patient

   1. is free of physical, psychological or other impairment that would prevent their ability to understand and comply with all study requirements.
   2. is willing and capable of providing Informed Consent to undergo study procedures.
   3. agrees to fully participate in all examinations, study requirements, follow-up visits and tests associated with this clinical study.
   4. lives close enough to the investigational site to facilitate the required in-person visits.

Exclusion:

1. Urologic conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to:

   1. Previous operative intervention for BPH
   2. Active urinary tract infection (may be treated and enrolled upon negative urine culture).
   3. Prostatitis: a history of any prostatitis within 2 years of enrollment.
   4. Cystolithiasis active within 90 days of enrollment
   5. artificial sphincters.
2. Bladder cancer: a history of treated bladder cancer of Stage T2 or higher, or a clinical suspicion of bladder cancer
3. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to:

   a. Unstable cardiovascular disease including: i. NYHA III/IV heart failure or LVEF < 40% ii. Uncontrolled arrhythmia iii. Stroke, TIA, thromboembolic event, myocardial infarction, unstable angina, percutaneous coronary intervention or any cardiac surgery within 90 days of enrollment iv. Uncontrolled hypertension b. Immunosuppression: Known immunosuppression, including but not limited to AIDS, immunosuppressive medication or current chemotherapy.

   c. Coagulopathy: Diagnosed disorder of blood clotting or bleeding diathesis. d. Transplant: History of any solid organ or hematologic transplant, or currently being evaluated for an organ transplant e. Active substance abuse: active alcoholism or

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Outcome | 30 days
  The safety endpoint for this study is a Composite Safety Endpoint (CSE) defined as the proportion of subjects with one or more device- or procedure-related serious adverse events (SAEs) through 30 days post-procedure.

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (2):
  - Brno University Hospital, Brno
  - Urologicka Klinika, Hradec Králové
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
- Pacifica Salud Hospital, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No